CLINICAL TRIAL: NCT05030896
Title: Clinical Application of Percutaneous Electrolysis in Female Soccer
Brief Title: Ultrasound-guided Percutaneous Electrolysis in Female Soccer With Soleus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Doctor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Female Soccer
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive EPM and they will perform exercise program during 1 month.
  Interventions: Other: Invasive treatment and exercise therapy
- Control group (Experimental): Participants will receive needling puncture and they will perform exercise program during 1 month.
  Interventions: Other: Invasive treatment and exercise therapy

INTERVENTIONS:
Other: Invasive treatment and exercise therapy — The subjects of experimental group will perform therapeutic exercise program and they will be receive Percutaneous Electrolysis therapy and the subjects of experimental group will perform the same exercise program and they will be receive only needling puncture

SUMMARY:
This study evaluates if the physiotherapy treatment based on combination of therapeutic exercise program and ultrasound-guided PNE on chronic soleous injuries may cause changes in pain, dorsal flexion of the ankle and muscle fatigue in female dance

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* having a soleus muscle injury
* chronic injury (> 3 meses)
* pain at stretch > 3 points measured by NRS

Exclusion Criteria:

* belenophobia
* other accuse injury
* lumbar back pathology

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Pain at palpation | From baseline measurement up to one month
  measured by numeric rate scale (0 no pain; 10 worst pain)
Pain at stretch | From baseline measurement up to one month
  measured by numeric rate scale (0 no pain; 10 worst pain)

SECONDARY OUTCOMES:
ankle dorsiflexion | From baseline measurement up to one month
  range of motion measured by goniometer (grade)
muscle fatigue | From baseline measurement up to one month
  measured by heel test: raise until muscle fatigue (repetitions)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain